CLINICAL TRIAL: NCT02803762
Title: A Phase 1, Open-Label Study to Investigate the Absorption, Metabolism, Excretion, and Mass Balance of [14C] Pacritinib Following a Single Oral Dose in Healthy Male Subjects
Brief Title: Investigate Absorption, Metabolism, Excretion, and Mass Balance of Pacritinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Collaborators: QPS-Qualitix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PAC102
Record Dates: First submitted 2016-05-03; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: ADME; Pacritinib
MeSH Terms: interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigational: [14C] Pacritinib (Experimental): All enrolled subjects are checked in the day before drug administration. Following at least a 10-hour fast (not including water), each subject will receive an oral dose of 400 mg [14C]pacritinib (containing 100 μCi radioactivity).
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib — 400 mg [14C]pacritinib (containing 100 μCi radioactivity) administered orally as a single dose following at least a 10-hour fast (not including water) on Day 1

SUMMARY:
This study is an open-label, absorption, metabolism, excretion, and mass balance study of 400 mg [14C]pacritinib (containing 100 μCi radioactivity) administered orally as a single dose to 6 healthy male subjects following at least a 10-hour fast (not including water) on Day 1.

DETAILED DESCRIPTION:
The present study is designed to investigate the absorption, metabolism, excretion as well as safety/tolerability of pacritinib following the administration of a single oral dose to healthy male volunteers. The pacritinib dose is administered with a [14C]-labeled form to enable detection and quantitation of dose-related material independent of possible biotransformation. The study design allows detection of potential human specific metabolites that have not been detected in the animal species. Subjects are confined at the clinical site from the time of Check-in until Day 14 post-dose, but may be discharged from the clinical site between Day 10 and 13 post-dose if study discharge criteria are met (i.e. completion of sufficient radioactivity excretion). All remaining subjects will be discharged from the clinical site on Day 14 post-dose irrespective of the study discharge criteria. The data obtained in this study will be used for the further clinical development of the compound.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking men between 18 and 55 years of age (inclusive)
* ECG within normal limits (according to the criteria used by QPS Netherlands BV including QTc interval (less than or equal to 450 m/sec)
* Normal vital signs measurements [defined as blood pressure (BP) between 90-140 mmHg systolic and 50-90 mmHg diastolic, resting heart rate (HR) between 40-100 beats/min, temperature (T) less than or equal to 37.6 degree C])
* Body mass index of 19.0-29.0 kg/m2 inclusive
* Negative history of drug abuse or alcoholism within 1 year prior to Day 1
* Negative tests on drug and alcohol screen at Screening and Check-in
* Negative hepatitis panel including hepatitis B-surface antigen HBsAg], hepatitis C antibody [anti-HCV] and negative human immunodeficiency virus antibody (HIV)
* No clinical laboratory value outside of the normal reference range unless deemed not clinically significant by the Investigator in consultation with the Sponsor
* Fertile male subjects and fertile female sexual partners of male subjects agree to use effective birth control methods throughout the entire study. Female partners of childbearing potential must use highly effective methods (defined as those resulting in a failure rate of <1% per year when used consistently and correctly). The contraceptive methods considered highly effective are intrauterine devices and hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices, or injections with prolonged release). Male subjects must use a condom with spermicide paste for the duration of the study and for 90 days after the EOS evaluation. When abstinence is used as a method of birth control, only true abstinence is acceptable, when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (calendar, ovulation, symptothermal, and post-ovulation methods) and withdrawal are not acceptable methods of contraception
* Agreement to not donate sperm throughout the entire study and for 3 months after the end of the study
* Willingness to comply with the protocol, including restrictions on diet, physical activity, and use of alcohol, medications, and other drugs during the study
* Comprehend and willingness to sign an approved informed consent form for the study
* At least one bowel movement a day

Exclusion Criteria:

* Participation in another radioactive clinical trial within the past 12 months
* Actively participating in an experimental therapy study or who have received experimental therapy within 90 days of Day 1
* Use of any other prescription medication within 21 days of Day 1, unless approved by Sponsor
* Use of over-the-counter (OTC) medications or nonprescription preparations (including vitamins, minerals and phytotherapeutic/herbal/plant-derived preparations) that is known to induce drug-metabolizing enzymes, including CYP450 enzymes within the 7 days preceding Day 1 (except for spermicidal/barrier contraceptive products and paracetamol)
* Consumption of alcoholic beverages within 72 hours prior to Check-in (Day -1)
* Consumption of grapefruit- and grapefruit-containing products within 7 days prior to Day 1
* Consumption of xanthine containing beverages such as coffee, including energy drinks containing caffeine or tea within 2 days of Day 1
* Clinically significant abnormal physical finding at Screening
* Any severe acute or chronic medical condition, psychiatric condition, or laboratory abnormality that in the Investigator's opinion may increase the risk associated with study participation or administration of study treatment, or interfere with the interpretation of study results (such as gastrointestinal surgical history (except appendectomy), ileus or obstructive uropathy)
* Diarrhea, nausea or vomiting within 7 days of Day 1
* History of additional risk factors for torsade de pointes (TdP) (e.g. heart failure, hypokalemia defined as serum potassium <3.0 mmol/L, family history of Long QT Syndrome)
* Any illness during the 4 weeks prior to Day 1, unless deemed NCS by the Principal Investigator
* Any history of severe allergic reaction (including drugs, food, insect bites, environmental allergens)
* Known history or presence of food allergies or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
* Any surgical procedures within 72 hours of Day 1
* Blood draws of more than 400 mL during the conduct of any clinical study within 90 days prior to Day 1
* Poor peripheral venous access
* Donation of blood 30 days prior to Screening through end of study
* Employment in a position that exposes the subject to radiation or requires that the subject's degree of radiation exposure be monitored (e.g. radiology technician)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) | 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose every 24 hours thereafter until Day 10, no later than Day 14
  The PK parameters for [14C] pacritinib will be derived by non-compartmental analysis of the plasma concentration-time profiles and the PK parameters for the metabolites will be calculated, as deemed appropriate, based on the results of quantitative profiling performed on selected plasma and pooled urine samples from individual subjects
The time to reach maximum plasma concentration (tmax) | 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose every 24 hours thereafter until Day 10, no later than Day 14
  The PK parameters for [14C] pacritinib will be derived by non-compartmental analysis of the plasma concentration-time profiles and the PK parameters for the metabolites will be calculated, as deemed appropriate, based on the results of quantitative profiling performed on selected plasma and pooled urine samples from individual subjects
The area under the plasma concentration-time curve from time zero to time of the last measured concentration above the limit of quantification (AUC0-t) | 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose every 24 hours thereafter until Day 10, no later than Day 14
  The PK parameters for [14C] pacritinib will be derived by non-compartmental analysis of the plasma concentration-time profiles and the PK parameters for the metabolites will be calculated, as deemed appropriate, based on the results of quantitative profiling performed on selected plasma and pooled urine samples from individual subjects
The area under the plasma concentration-time curve from time zero to 48 hours (AUC0- 48h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose every 24 hours thereafter until Day 10, no later than Day 14
  The PK parameters for [14C] pacritinib will be derived by non-compartmental analysis of the plasma concentration-time profiles and the PK parameters for the metabolites will be calculated, as deemed appropriate, based on the results of quantitative profiling performed on selected plasma and pooled urine samples from individual subjects
The area under the plasma concentration-time curve from zero to infinity (AUC0-∞) | 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose every 24 hours thereafter until Day 10, no later than Day 14
  0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose every 24 hours thereafter until Day 10, no later than Day 14

SECONDARY OUTCOMES:
Treatment-emergent adverse events (AEs) and serious adverse events (SAEs), vital Signs, PE, clinical laboratory valuations, and ECGs | Day 1 through Day 42
  Evaluate Safety and tolerability of a single oral dose of 400 mg [14C]pacritinib in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Khalid A Elaziz, MBBS, MD, Principal Investigator — QPS Netherlands BV
Locations (1):
- QPS Netherlands B.V., Groningen, Netherlands